CLINICAL TRIAL: NCT06940271
Title: RAP: Prospective Pragmatic Multi-Site Trial Evaluating the Feasibility and Effect of Wrapping the Cavernous Nerves With a Novel Multi-Layer Perinatal Tissue Allograft During Prostatectomy
Brief Title: Feasibility and Effect of Wrapping Nerves With a Multi-Layer Perinatal Tissue Allograft During Prostatectomy
Acronym: RAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MC240501; NCI-2025-02552 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-013215 (Other: Mayo Clinic Institutional Review Board); MC240501 (Other: Mayo Clinic)
Record Dates: First submitted 2025-04-15; First posted 2025-04-23 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Localized Prostate Carcinoma; Stage I Prostate Cancer AJCC v8; Stage II Prostate Cancer AJCC v8; Stage III Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Transplantation, Homologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (MLG-Complete allograft) (Experimental): Patients undergo placement of MLG-Complete allograft to nerve bundles over 5 minutes during standard of care nerve-sparing RARP.
  Interventions: Procedure: Allografting; Other: Survey Administration

INTERVENTIONS:
Procedure: Allografting — Undergo placement of MLG-Complete allograft
  Other Names: allograft
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial studies whether a new multi-layer perinatal tissue allograft, MLG-Complete (Trademark), can be used to improve complications after nerve-sparing robot-assisted radical prostatectomy (RARP) in patients with prostate cancer that has not spread to other parts of the body (localized). Two major complications that can happen after complete surgical removal of the prostate (radical prostatectomy) include erectile dysfunction and urinary incontinence, both of which greatly affect a patient's quality of life and social well-being. The goal of nerve-sparing radical prostatectomy is to preserve erectile and urinary function, but damage to the surrounding nerves and blood vessels can still occur causing the patient to experience the complications. An allograft is the transplant of an organ, tissue, or cells from one individual to another individual of the same species who is not an identical twin. The MLG-Complete allograft is made up of perinatal tissue and is placed on the nerve bundles during a nerve-sparing RARP. It is meant to serve as a barrier and provide coverage to the nerve bundles from the surrounding environment, which may improve post-nerve-sparing RARP complications.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects with age ≥ 45
* Primary diagnosis of prostate cancer selected for surgical intervention (radical prostatectomy)
* Primary diagnosis of organ confined (i.e. localized) untreated prostate cancer
* Planned elective radical prostatectomy with bilateral nerve sparing technique
* Negative urinalysis within 30 days prior to date of surgery
* Patient has no erectile dysfunction (SHIM score ≥ 19) at the time of consultation
* Willing to comply with instruction of the investigator
* Willing to comply with follow-up surveys
* Ability to provide written consent
* Negative urinary tract infection at the time of consultation
* Interest in penetrative sexual intercourse

Exclusion Criteria:

* High-risk cancer planned for neoadjuvant therapy, full or partial excision of neurovascular bundles
* Unable to comply with learning and documenting penile rehabilitation, including oral 5-phosphodiesterase inhibitor use, vacuum pump therapy use, and/or injectable medications
* History of >14 days treatment with immunosuppressants (including systemic corticosteroids), cytotoxic chemotherapy within one month prior to initial screening, or who receive such medications during the screening period
* Prior hormonal therapy such as Lupron or oral anti-androgens
* Poor urinary control at baseline requiring the use of pads for leakage
* Previous history of pelvic radiation
* Previous history of simple prostatectomy or transurethral prostate surgery
* Patients with obesity defined as body mass index (BMI) > 40 kg/m^2
* History of open pelvic surgery ≤ 5 prior to registration (except for hernia repair)
* Scheduled to undergo chemotherapy, radiation, hormone therapy, or open surgery during the study period
* Any neurologic disorder or psychiatric disorder that might confound postsurgical assessments
* Has any condition(s) which seriously compromises the subject's ability to participate in this study, sign consent, or has a known history of poor adherence with medical treatment
* In the opinion of the principal investigator (PI), has a history of drug or alcohol abuse ≤ 12 months prior to registration
* Allergic to aminoglycoside antibiotics (such as gentamicin and/or streptomycin)
* Received administration of an investigational drug within 30 days prior to registration, and/or has planned administration of another investigational product or procedure during participation in this study

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2030-07-30 (Estimated); Study Completion 2030-07-30 (Estimated)

PRIMARY OUTCOMES:
Ability to place MLG-Complete allograft without lengthening operative time (Feasibility) | Baseline [time of robot-assisted radical prostatectomy (RARP)]
  Feasibility is defined as the overall technical ability to place the MLG-Complete allograft in included patients without significantly lengthening operative time. This will be defined by a yes/no evaluation by the surgeon.
Incidence of serious adverse events related to graft placement | Up to 6 weeks post-RARP
  Will be assessed according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
Average time for return of potency | At 6-weeks and 3-, 6-, and 12-months post RARP
  Will be defined as the ability to achieve an erection sufficient for intercourse for at least 50% of the time or at least 50% rigidity post RARP. Will be assessed using the Sexual Health Inventory for Men (SHIM) and patient-reported history. The SHIM is a five-question instrument with a score of 1-25 points. A higher score generally indicates greater ability to achieve an erection.
Average time for return to continence | At 6-weeks and 3-, 6-, and 12-months post-RARP
  Return to continence will be defined as use of =< 1 pad post-RARP.
Change in SHIM | At baseline, 6-weeks post-RARP, and 3-, 6-, and 12-months post-RARP
  Sexual Health Inventory for Men (SHIM) scores will be collected at study enrollment, 6 weeks, 3 months, 6 month, and 12 months. The SHIM consists of five questions that explore aspects of erectile function. Scores range from 1-25. A score of 20 or higher indicates a normal degree of erectile functioning. Lower scores (10 or less) indicate moderate to severe erectile dysfunction (ED).
Change in AUASS | At baseline, 6-weeks post-RARP, and 3-, 6-, and 12-months post-RARP
  The American Urological Association Symptom Score (AUASS) consists of 5 questions related to urological symptoms over the past month. Questions are answered on a scale of 0-5 where 0=not at all and 5=almost always and one question related to nighttime urination (times per night average over the past month). A lower overall score indicates lesser urological symptoms.
Change in Quality of Life - AUASS survey | At baseline, 6-weeks post-RARP, and 3-, 6-, and 12-months post-RARP
  Assessed with a single survey question answered on a scale of 0-6 where 0=delighted and 6=terrible.
Change in ICIQ-UI | At baseline, 6-weeks post-RARP, and 3-, 6-, and 12-months post-RARP
  The International Consultation on Incontinence Questionnaire: Short Form for Urinary Incontinence (ICIQ-UI) is a 4-item questionnaire related to urine incontinence over the past 4 weeks. A higher summary scores indicates worse incontinence.
Change in QoL - EPIC-26 | At baseline, 6-weeks post-RARP, and 3-, 6-, and 12-months post-RARP
  The Expanded Prostate Cancer Index Composite (EPIC-26) is a 26-item questionnaire related to Quality of Life issues in patients with Prostate Cancer. The survey consists of 26 items under 5 domains: urinary incontinence, urinary irritative/obstructive, bowel, sexual, and hormonal.
Cost/value analysis | Up to 12 months post-RARP
  Costs of prescription [Oral Phosphodiesterase 5 Inhibitor (PDE-5i), Intracavernosal injection, Alprostadil urethral suppository) or future surgery (inflatable penile prosthesis] will be recorded.
Unplanned interactions with the healthcare team | Up to 12 weeks
  The proportion of patients with an unplanned phone call, portal message, or unscheduled clinic, emergency room, or urgent care visit will be computed and presented. The total number of unplanned phone calls, portal messages, or health care visits will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Ram A. Pathak, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials